CLINICAL TRIAL: NCT06886893
Title: Optical Coherence Tomography Data As a Prognostic Indicator in Retinal Vein Occlusion
Brief Title: Optical Coherence Tomography in Retinal Vein Occlusion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mayar Adel Francis, resident at the ophtalmology department, Assiut University
Other Study IDs: OCT in retinal vein occlusion
Record Dates: First submitted 2025-03-15; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Optical Coherence Tomography (OCT)
Keywords: OCT; retinal vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with branch or central RVO, macular edema confirmed by OCT, and no prior RVO in the affected: Adults aged 18 years or older.
  Patients diagnosed with branch or central retinal vein occlusion.
  Patients with macular edema confirmed by OCT due to vein occlusion.
  Patients with no prior history of RVO in the affected eye.

SUMMARY:
This study aims to evaluate how optical coherence tomography (OCT) can help predict outcomes in patients with retinal vein occlusion (RVO), a condition that affects blood flow in the retina. RVO can cause macular edema, which is swelling in the part of the eye responsible for central vision. The study will use OCT scans to assess changes in the retina and how these changes relate to vision improvement over time.

DETAILED DESCRIPTION:
Objectives Evaluate how OCT data can predict visual outcomes by analyzing retinal changes and macular edema characteristics.

Assess the correlation between baseline OCT biomarkers and visual acuity improvements over time.

Study Design Type: Cross-sectional study.

Setting: Conducted at several eye care centers in Egypt.

Participants Inclusion Criteria: Adults with branch or central RVO, macular edema confirmed by OCT, and no prior RVO in the affected eye.

Exclusion Criteria: Other retinal diseases, recent intraocular surgery, or significant media opacities.

Procedures Informed Consent and History Taking.

Ophthalmologic Examination: Includes BCVA, IOP, slit-lamp biomicroscopy, and fundus examination.

OCT Imaging: Using NIDEK RS-330 Retina scan duo 2 (SD-OCT) to assess macular changes.

OCT Image Evaluation: Classification of macular edema types and assessment of biomarkers like subretinal fluid and cystoid changes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.

Patients diagnosed with branch or central retinal vein occlusion.

Patients with macular edema confirmed by OCT due to vein occlusion.

Patients with no prior history of RVO in the affected eye.

Exclusion Criteria:

* Presence of other retinal diseases that could affect OCT interpretation (e.g., diabetic retinopathy, age-related macular degeneration).

History of intraocular surgery within the last three months.

Presence of significant media opacities (e.g., dense cataract, vitreous hemorrhage) that interfere with OCT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with retinal vein occlusion (RVO), a condition that affects blood flow in the retina. RVO can cause macular edema, which is swelling in the part of the eye responsible for central vision. Adults aged 18 or older with branch or central retinal vein occlusion. Patients must have macular edema confirmed by OCT and no previous RVO in the affected eye.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
changes in OCT biomarkers and visual acuity post-treatment. | 6 months
  Correlation between baseline OCT biomarkers and visual acuity at presentation after 1, 3, and 6 months post-treatment.

IPD SHARING:
Plan to Share IPD: No